CLINICAL TRIAL: NCT06523192
Title: The English Version of the Drug Hypersensitivity Quality of Life Questionnaire: Validity and Reliability in the British Population.
Brief Title: Validation of the English Version of the Drug Hypersensitivity Quality of Life Questionnaire
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 151058
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Drug Hypersensitivity; Quality of Life
MeSH Terms: conditions — Drug Hypersensitivity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — No intervention

SUMMARY:
We aim to validate the English (UK) translation of the DrHy-Q, and test its reliability in the UK population. This will facilitate for the subsequent economical evaluation of penicillin allergy delabelling.

This research project is part of an MSc in Allergy undertaken by the principal applicant, Dr Patricia Romero, supervised through Imperial College London.

Target population are patients with a drug allergy diagnosed by an Allergist prospectively at the Drug Allergy Clinic.

Is the English version of the Drug Hypersensitivity Quality of Life Questionnaire suitable to be used in the UK population?

ELIGIBILITY:
Inclusion Criteria:

* • Age >18 years

  * Ability to read English and consent.
  * Confirmed diagnosis of a drug hypersensitivity reaction.
  * Written informed consent

Exclusion Criteria:

* • < 18y/o.

  * Not able to read English. No mental capacity to consent or unwilling to consent.
  * Unconfirmed diagnosis of a drug hypersensitivity reaction.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Our target population are patients with diagnosed drug allergy.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Validation of the English version of the Drug Hypersensitivity Questionnaire | March 2023 May 2024
  Reliability and validity

CONTACTS AND LOCATIONS:
Locations (1):
- UNiversity Hospitals Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No